CLINICAL TRIAL: NCT01202500
Title: Multicentre, Randomised Study to Determine the Relative Efficacy of Two Therapeutic Strategies in the Treatment of Children With Congenital Toxoplasmosis
Brief Title: Assessment of Two Therapeutic Strategies in the Treatment of Children With Congenital Toxoplasmosis
Acronym: TOSCANE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Fansidar marketing discontinued
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-016528-30
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Congenital Toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 months (Other)
  Interventions: Procedure: registered length of treatment
- 3 months (Experimental)
  Interventions: Procedure: reducing treatment to 3 months

INTERVENTIONS:
Procedure: reducing treatment to 3 months — The treatment will be stopped after 3 months
  Arms: 3 months
Procedure: registered length of treatment — The treatment procedure will follow the actual recommandation
  Arms: 12 months

SUMMARY:
Toxoplasmosis is a benign disease in healthy adults, but can be serious in the case of contamination during pregnancy: the parasite can pass through the placental barrier and infect the foetus. The severity of congenital infection varies, but in France, where maternal seroconversions during pregnancy are treated, the manifestations of the disease are often infraclinical at birth and only appear during the first years of life in the form of retinochoroiditis. In order to prevent long-term sequellae, children with confirmed congenital toxoplasmosis (TC) are treated with pyrimethamine combined with either sulfadiazine or sulfadoxine (Fansidar®). The relative efficacy of these two combinations has not yet been evaluated. Moreover, there is no consensus about the duration of the treatment, which varies, in France, from 12 to 24 months depending on the centre. Compared with the duration of parasitaemia in non-treated children, which can persist for up to 4 weeks, these treatments are very long. They are also far longer than the 3 months of treatment, which is in accordance with the World Health Organization (WHO) recommendations, given in Denmark to infants identified as being infected with the parasite during neonatal screening. A one-year treatment was developed in the United States, but it mainly concerns only symptomatic children, given the absence of generalised screening in the United States of America (USA). We have no arguments to justify the use of treatments lasting one year or more in children with asymptomatic or mildly-symptomatic TC. As these treatments carry certain risks, which may be severe, notably with regard to haematological or skin conditions, they have to be supervised closely with biological tests, which adds further constraints for both the children and their parents and increases the cost to health care systems.

ELIGIBILITY:
Inclusion Criteria:

Children meeting the following criteria can be included:

* Non-severe congenital toxoplasmosis diagnosed in utero or in the first 3 months of life, whether or not in utero treatment was given
* Treated for 3 months with pyrimethamine combined with sulfamides.
* age from 3 to 6 months (> 2 months and < 7 months)

Diagnostic criteria for congenital toxoplasmosis:

* antenatal period: positive Polymerase Chain Reaction (PCR) on the amniotic fluid or positive mouse inoculation for the amniotic fluid
* postnatal period: presence of specific Immunoglobuline M (IgM) and/or Immunoglobuline A (IgA), positive Western Blot Chemistry (WBC), increase in Immunoglobuline G (IgG).

Severe congenital toxoplasmosis is defined by the presence at birth of at least one of the following signs: > or egal 3 cerebral calcifications, hydrocephaly, microcephaly, convulsions, microphtalmy.

Informed consent must be provided by both parents.

Exclusion Criteria:

Children with the following cannot be included:

* a severe form of congenital toxoplasmosis
* inflammatory retinal disease at inclusion or in whom the treatment is contra-indicated (history of hypersensitivity to one of the components, severe renal or hepatic insufficiency, a history of hepatitis linked to treatment with Fansidar®).

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
episode of retinochoroiditis | 2 years
  Time to the onset of a first episode of retinochoroiditis in the two years of the study (or the onset of a new episode in a child known to already have had at least one lesion), evaluated on a fundus examination using RetCam®.

CONTACTS AND LOCATIONS:
Overall Officials: Christine BINQUET, MD, Study Director — CHU Dijon
Locations (1):
- Hôpital d'Enfants Armand Trousseau, Paris, France